CLINICAL TRIAL: NCT02582918
Title: Comparative Effectiveness Trial of Care Delivery Strategies for HCC Screening Process Completion
Brief Title: Texas Hepatocellular Carcinoma Consortium (THCCC) Project 5
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Parkland Health and Hospital System (Other); Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Amit Singal, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 062015-054
Record Dates: First submitted 2015-10-13; First posted 2015-10-21 (Estimated); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Carcinoma, Hepatocellular; Liver Neoplasms
Keywords: Randomized Controlled Trial; Mass Screening
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Patient Education as Topic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Usual Care (No Intervention): Usual care with opportunistic visit-based HCC surveillance.
- Group 2: Patient Education and Patient Navigation Services (Experimental): Mailed HCC surveillance outreach with patient education and patient navigation services.
  Interventions: Behavioral: Outreach with patient education and patient navigation services

INTERVENTIONS:
Behavioral: Outreach with patient education and patient navigation services — * Outreach invitations include number to call for more information about scheduling an ultrasound and alpha fetoprotein (AFP) blood test.
  * Patients receive up to three phone calls 2-4 weeks after invitations and a reminder call 5-7 business days before appointments.
  * If results are normal, the patient is invited to repeat screening in 6 months.
  * If suspicious mass on ultrasound or abnormal AFP level, the patient is referred for follow-up testing with triple-phase CT scan or MRI.
  * If CT/MRI is unremarkable, the patient is referred back for routine screening.
  * If HCC is confirmed, the patient and their primary care provider will be contacted with the results.
  * All patients diagnosed with HCC will be seen in the multi-disciplinary HCC clinic.
  Arms: Group 2: Patient Education and Patient Navigation Services

SUMMARY:
Project 5 of the Texas HCC Consortium (THCCC) is a comparative effectiveness pragmatic randomized control trial (RCT) of outreach strategies to increase hepatocellular cancer (HCC) surveillance process completion among a socioeconomically and racially diverse cohort of Texans with cirrhosis. Through this project the investigators will implement and evaluate system-level mailed outreach interventions to identity at-risk patients with cirrhosis, promote HCC surveillance, and ensure timely follow-up of tests at UT Southwestern (UTSW) Medical Center, Parkland Health and Hospital System (PHHS), and the Houston Veterans Affairs (VA) Medical Center. The study population will include adult patients with documented or unrecognized cirrhosis and at least one outpatient clinic visit in year prior to randomization. Patients will be identified using an EMR-enabled case identification algorithm. The investigators will randomize 3000 patients (1500 per arm) identified by this algorithm to: usual care, with opportunistic visit-based HCC surveillance (Group 1); or, mailed HCC surveillance outreach with patient education and patient navigation services (Group 2).

DETAILED DESCRIPTION:
Hepatocellular cancer (HCC) is the most common (≥ 95%) of liver cancers. HCC is also the fastest rising cause of cancer-related deaths in the U.S. HCC is particularly important for Texas residents. Texas has the second highest death rate from HCC in the nation. The 5-year HCC survival remains low (10-15%) and most patients get diagnosed at late stages. Texas residents notably Hispanics and African Americans are greatly affected with established HCC risk factors including hepatitis C virus, hepatitis B virus and alcoholic liver disease. Furthermore, emerging HCC risk factors, specifically the metabolic syndrome and non-alcoholic fatty liver disease (NAFLD), are exceptionally common in Texans.

The goal of the Texas Hepatocellular Carcinoma Consortium (THCCC) is to reduce the death and suffering related to liver cancer in Texas and the world through five research projects.

This protocol outlines Project 5 of the THCCC which is a comparative effectiveness randomized controlled trial of strategies to increase HCC surveillance. This is the first multi-center outreach intervention aimed at improving surveillance process completion among at-risk patients with cirrhosis.

This study is based at 3 health systems in Texas: UT Southwestern (UTSW) Medical Center, Parkland Health and Hospital System (PHHS), and the Houston Veterans Affairs (VA) Medical Center. Across these 3 sites, we will implement and evaluate system-level mailed outreach interventions to identity at-risk patients with cirrhosis, promote HCC surveillance, and ensure timely follow-up of tests. This study uses an EMR-enabled case-finding algorithm to identify patients with documented cirrhosis, using ICD-9 codes, and those with unrecognized cirrhosis, using laboratory data.

Over 3000 patients identified by this algorithm will be randomized to:

* Group 1: Usual care with opportunistic visit-based HCC surveillance.
* Group 2: Mailed HCC surveillance outreach with patient education and patient navigation services.

The Specific Aims are:

* Aim 1: Compare the clinical effectiveness of the intervention strategies to increase completion of the HCC surveillance process.
* Aim 2: Compare patient-reported satisfaction and acceptability of the HCC surveillance strategies.
* Aim 3: Evaluate whether intervention effects are moderated by patient sex, race/ethnicity, socioeconomic status, health care utilization, and documented vs. unrecognized cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>21 years old)
* Documented cirrhosis
* Unrecognized cirrhosis
* An outpatient visit in year prior to randomization
* English or Spanish speaking

Exclusion Criteria:

* History of HCC
* History of liver transplantation
* Child Pugh C cirrhosis
* Significant comorbid conditions with life expectancy < 1 year, (e.g., extrahepatic malignancy)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2871 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Completion of HCC surveillance process | 3 years post randomization
  Ascertained through EMR.
  HCC surveillance process completion will be defined as:
  * normal ultrasound and AFP every 6 ± 1 months for two consecutive years,
  * abnormal ultrasound or AFP ≥20 ng/mL and follow-up diagnostic CT or MRI without HCC, then appropriate surveillance as indicated for total of 2 years, or
  * abnormal ultrasound or AFP, HCC detected on CT/MRI, and timely HCC treatment consultation.
  Effective surveillance requires repeat testing every 6 months in patients with normal tests to maximize sensitivity while minimizing patient burden.
  Patients with abnormal surveillance tests (i.e. liver mass on ultrasound or AFP ≥20 ng/mL) require 4-phase CT or MRI within 3 months, with a 3-month cut-off based on HCC tumor doubling time.
  Patients with non-contrast imaging, two-phase CT, or imaging > 3 months after abnormal tests will be coded as failure.
  Likewise, patients with HCC confirmed on CT/MRI will need HCC-directed treatment within 3 months.
Patient satisfaction and acceptability | 3 years post randomization
  Assessed by 15-20 minute telephone semi-structured interviews.
  Patients will be called >24 months post-randomization to ensure interviews do not interfere with likelihood of surveillance process completion.
  The investigators will interview 30 completers and 30 non-completers from each group at each site (540 total).
  The investigators will stratify sampling to include both patients with documented cirrhosis and unrecognized cirrhosis. Likert scale items will assess reactions:
  * Participants were confused why they were referred for HCC screening
  * Participants were not given enough information to make a decision
  * Participants don't want to know if they have HCC
  * Information about HCC was new and items assessing if invitations included more, right amount, or not enough information as the participants would like.
  Interviews will also assess what HCC testing (if any) patients think they should have.

SECONDARY OUTCOMES:
Early HCC | 3 years post randomization
  HCC will be defined by AASLD criteria and staged by Barcelona Clinic Liver Cancer (BCLC) system.
  Tumors >1 cm can be diagnosed if CT/MRI shows characteristic findings (arterial enhancement and delayed washout).
  Biopsy may be needed if imaging is not diagnostic.
  Early HCC will be defined as BCLC stage A tumors that are amenable to curative therapy.
  HCC diagnoses and stage will be ascertained from EMR data and confirmed by site investigators.
One-time Screening | Outcomes will be adjudicated 6 months after randomization.
  Defined as the proportion of patients completing HCC screening within 6 months of randomization.
Repeat Screening | Outcomes will be adjudicated 12 months after randomization.
  Defined as the proportion of patients completing HCC screening every 6 months within 12 months of randomization. Patients will be categorized as completed all screening (2 screening in 12 months), some screening (1 screening in 12 months), or no screening (0 screening in 12 months).

CONTACTS AND LOCATIONS:
Overall Officials: Amit G Singal, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Derived] Singal AG, Daher D, Narasimman M, Yekkaluri S, Liu Y, Cerda V, Banala C, Khan A, Lee M, Seif El Dahan K, Murphy CC, Kramer JR, Hernaez R. Benefits and harms of hepatocellular carcinoma screening outreach in patients with cirrhosis: a multicenter randomized clinical trial. J Natl Cancer Inst. 2025 Feb 1;117(2):262-269. doi: 10.1093/jnci/djae228. PMID 39288308
- [Derived] Singal AG, Narasimman M, Daher D, Yekkaluri S, Liu Y, Lee M, Cerda V, Khan A, Seif El Dahan K, Kramer J, Gopal P, Murphy C, Hernaez R. Effectiveness of mailed outreach and patient navigation to promote HCC screening process completion: a multicentre pragmatic randomised clinical trial. Gut. 2024 Nov 11;73(12):2037-2044. doi: 10.1136/gutjnl-2024-332508. PMID 38839269
- [Derived] Singal AG, Reddy S, Radadiya Aka Patel H, Villarreal D, Khan A, Liu Y, Cerda V, Rich NE, Murphy CC, Tiro JA, Kramer JR, Hernaez R. Multicenter Randomized Clinical Trial of a Mailed Outreach Strategy for Hepatocellular Carcinoma Surveillance. Clin Gastroenterol Hepatol. 2022 Dec;20(12):2818-2825.e1. doi: 10.1016/j.cgh.2021.12.014. Epub 2021 Dec 10. PMID 34902568